CLINICAL TRIAL: NCT00466544
Title: Randomized Controlled Study of Plasmaknife Tonsillectomy Versus Monopolar Tonsillectomy
Acronym: jPK
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Children's Hospital of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 036706MP4F
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-03

CONDITIONS: Obstructive Tonsillar Hypertrophy; Tonsillitis
Keywords: Chronic tonsillitis; Recurrent tonsillitis
MeSH Terms: conditions — Tonsillitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Plasmaknife
Device: Monopolar

SUMMARY:
Study objective is to provide prospective randomized controlled data on pediatric pain levels found in PlasmaKnife tonsillectomy and monopolar tonsillectomy.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled study to compare the efficacy of the Gyrus ACMI PlasmaKnife™ electrosurgical device used with the Gyrus ACMI Workstation versus monopolar electrosurgical device (i.e. Bovie®) for tonsillectomy.

The primary outcome will study the potential for reduced post-operative pain when the PlasmaKnife is used for tonsillectomy compared to a monopolar device. Secondary outcomes such as return to normal diet and activity as well as a range of complications including primary and secondary bleeding will be included in the study.

The study will involve approximately 100 patients at Children's Hospital of Michigan that meet the criteria for tonsillectomy (with or without adenoidectomy) for infected tonsils or airway obstruction.

The study will be documented through the use of Case Report Forms.

ELIGIBILITY:
Inclusion Criteria:

* Patient should be between the ages of 4 and 16 years old inclusive.
* Patient should meet criteria for tonsillectomy.
* Patient's guardian able and willing to complete patient diary and keep to the follow-up visit.
* Guardian able to understand English (written and oral).

Exclusion Criteria:

* Patient that has active medical implant(s) such as pacemaker, cochlear implant, etc.
* Patient has abnormal blood coagulation, history of easy bruising, bleeding disorders or uses anti-coagulants.
* Morbidly obese children (calculated BMI over 39)
* Patient that has history of malignancy or acute peritonsillar abscess
* Patient has Sickle Cell disease or is immunocompromised.
* Patient is pregnant or lactating.
* Active infection with fever greater than 101.5 degrees F.
* History of heart disease, diabetes or hypertension (with systolic blood pressure > 160 mmHg).
* Craniofacial anomaly.
* Biopsy of tonsil needed to rule out neoplasm.

Ages: 4 Years to 16 Years | Sex: All
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2007-05

PRIMARY OUTCOMES:
pain

SECONDARY OUTCOMES:
return to normal activity
return to normal diet
medication dose taken

CONTACTS AND LOCATIONS:
Overall Officials: David Madgy, Principal Investigator — Detroit Children's Hospital
Locations (1):
- Detroit Children's Hospital, Detroit, Michigan, United States